CLINICAL TRIAL: NCT06817681
Title: The Effect of Exercise-Induced Lactate on BDNF and Cognition
Brief Title: Exercise-Induced Lactate and Cognitive Function (ExLBC)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Jeremy Walsh, Assistant Professor, McMaster University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: ExLBC
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-08

CONDITIONS: Cognition; Sodium Bicarbonate; Lactate; Exercise
Keywords: Lactate; Sodium Bicarbonate; NaHCO3; Cognition; Executive Function; Acute Exercise
MeSH Terms: conditions — Motor Activity | interventions — Sodium Bicarbonate; Sodium Chloride; Sodium Chloride, Dietary

STUDY DESIGN:
Intervention Model Description: A randomized double-blind placebo-controlled crossover design will be used to test 2 conditions. Participants will ingest gelatin capsules containing: 1) 0.4 g/kg body weight of sodium bicarbonate (NaHCO3); or 2) 0.4 g/kg body weight of sodium chloride (NaCl) (placebo supplement).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Single dose of a placebo supplement (0.4 g/kg body weight of sodium chloride gelatin capsules).
  Interventions: Other: Placebo (Sodium Chloride)
- Sodium bicarbonate (NaHCO3) (Experimental): Single dose of sodium bicarbonate supplement (0.4 g/kg body weight of NaHCO3 gelatin capsules).
  Interventions: Dietary Supplement: Sodium Bicarbonate (NaHCO3)

INTERVENTIONS:
Dietary Supplement: Sodium Bicarbonate (NaHCO3) — Ingestion of gelatin capsules containing 0.4 g/kg body weight of sodium bicarbonate (NaHCO3) followed by 90 minutes of rest. Continuous high intensity cycling to be performed following 90-minute resting measures.
  Other Names: Baking Soda
  Arms: Sodium bicarbonate (NaHCO3)
Other: Placebo (Sodium Chloride) — Ingestion of gelatin capsules containing 0.4 g/kg body weight of sodium chloride (NaCl) followed by 90 minutes of rest. Continuous high intensity cycling to be performed following 90-minute resting measures.
  Other Names: Table Salt
  Arms: Placebo

SUMMARY:
A single bout of exercise can rapidly improve cognitive functions including memory, attention, and executive functions, which help us navigate through everyday life. However, we do not fully understand the mechanism behind this process. A promising candidate mechanism is lactate, which was previously considered merely a waste product of our muscles during exercise. It is now recognized as an important molecule that is used by the brain as an energy source. Studies have shown that increases in lactate during exercise are positively related to improved cognitive function after completion of exercise. Another potential mechanism involves the increase in neurotrophins such as brain-derived neurotrophic factor (BDNF) following exercise. The increase in lactate and BDNF during exercise may be connected to cause these cognitive improvements.

However, because lactate increases with higher exercise intensities, we currently do not know how lactate specifically impacts brain health. To address this, muscle and blood lactate concentrations can be experimentally manipulated during exercise using sodium bicarbonate (NaHCO3) supplementation and will allow us to explore how lactate specifically affects brain function.

The purpose of this project is to investigate the effect of exercise-induced lactate on BDNF and cognition following oral NaHCO3 supplementation in young adults. We hypothesize that BDNF levels will be higher, and cognition will be improved in executive function, visuospatial memory, and working memory in the NaHCO3 condition due to higher plasma lactate during exercise compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-35 years old.
* Perform ≥150 minutes of moderate-to-vigorous aerobic activity per week.

Exclusion Criteria:

* Diagnosis of Type 2 Diabetes.
* Presence of hypoglycaemia.
* History of concussion(s) with persistent symptoms.
* History of mental health conditions.
* History of cardiovascular events requiring hospitalization (e.g., heart attack).
* Pre-existing injuries that prevent completion of aerobic exercise.
* Presence of colour-blindness.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-02-10 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function (Executive Function) | 3-hour
  The Stroop Task will be used to measure executive function (selective attention and inhibitory control).

SECONDARY OUTCOMES:
Cognitive Function (Working Memory) | 3-hour
  The N-Back Test will be used to assess working memory.
Cognitive Function (Visuospatial Memory) | 3-hour
  The Spatial Span Test will be used to assess visuospatial memory.
Blood Lactate | 3-hour
  Venous blood samples will be obtained via intravenous catheter.
Sodium Bicarbonate (NaHCO3) | 3-hour
  Venous blood samples will be obtained via intravenous catheter.
Blood pH | 3-hour
  Venous blood samples will be obtained via intravenous catheter.
Brain-Derived Neurotrophic Factor (BDNF) | 3-hour
  Serum and plasma BDNF measured in venous blood samples will be obtained via intravenous catheter.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy J Walsh, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share individual patient data (de-identified) with researchers upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 12 months and ending 36 months following article publication.
Access Criteria: Anyone who wishes to access the data.